CLINICAL TRIAL: NCT05634863
Title: The Role of an Implantable Doppler Vascular Monitoring Device in Kidney Transplant Patients: a Feasibility Randomised Controlled Trial With an Embedded Qualitative Study.
Brief Title: CONtinuous Implantable DOppler Probe Monitoring in Renal Transplantation
Acronym: CONDOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21/SUR/626
Record Dates: First submitted 2022-02-01; First posted 2022-12-02 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Renal Artery Complications; Renal Vein Thrombosis
Keywords: Implantable Doppler probe; Renal vein thrombosis; Renal artery complications

STUDY DESIGN:
Intervention Model Description: Intervention group: kidney transplant patients with the vascular monitoring device):
  The kidney transplant patients will receive the Implantable continuous vascular monitoring device surveillance for the first 72 hours in addition to the standard care clinical observation as part of their postoperative care.
  Control group (kidney transplant patients with standard care clinical observation):
  The kidney transplant patients will receive the standard care clinical observation as part of their postoperative care.
  The results of the study will be determined by comparing the surgical outcomes in both the intervention and control group.
Masking Description: Blinding of the participants (kidney transplant patients) to the outcome of the randomisation will not be possible due to the nature of the intervention. Similarly, the healthcare professionals (clinicians and nurses) taking care of the patients and collecting the data postoperatively cannot be blinded. However, the Southwest transplant team acts in the best interest of the kidney transplant patients and declares no conflict of interest with the device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KIDNEY TRANSPLANT PATIENTS WITH THE IMPLANTABLE CONTINUOUS VASCULAR MONITORING DEVICE (Experimental): The intervention that is intended to be investigated is the implantable vascular monitoring device manufactured by COOK Medical Company. Its principle intended use is continuous monitoring of the graft perfusion (i.e. transplanted kidney) for the first 72 hours postoperatively. The kidney transplant patients in the intervention group will receive implantable continuous vascular monitoring device surveillance for the first 72 hours in addition to the standard care clinical observation as part of their postoperative care. The intervention will be removed after 72 hours postoperatively.
  Interventions: Device: Implantable Doppler probe manufactured by COOK Medical Company.
- KIDNEY TRANSPLANT PATIENTS WITH STANDARD CARE CLINICAL OBSERVATION (No Intervention): The kidney transplant patients in this group will receive the standard care clinical observation as part of their postoperative care. Their graft will be monitored postoperatively by the standard care clinical observation as per the NHS protocol.

INTERVENTIONS:
Device: Implantable Doppler probe manufactured by COOK Medical Company. — The continuous audible Doppler signals produced by the monitoring device represent the blood flowing in the renal artery. This is an indicator of graft perfusion. Cessation of audible Doppler signals is the key that may suggest hampered blood flow due to vascular complications. In the intervention group, the monitoring device will be used as an added mechanism to monitor graft perfusion.
  Arms: KIDNEY TRANSPLANT PATIENTS WITH THE IMPLANTABLE CONTINUOUS VASCULAR MONITORING DEVICE

SUMMARY:
INTRODUCTION Vascular complications in kidney transplantation constitute one-third of the early graft loss (EGL) that can be prevented by timely diagnosed cases. A vascular monitoring device may have a possible role in the early identification of graft hypoperfusion critical to reducing graft loss.

AIM To evaluate the feasibility of an Implantable Doppler probe as a vascular monitoring device in kidney transplant patients and by obtaining the vital information, inform the protocol development of a definitive RCT.

METHODS AND ANALYSIS A mixed-method research design is selected. The quantitative study will comprise a feasibility RCT (fRCT) that will compare demographical characteristics and surgical outcomes of patients that will undergo kidney transplant surgery with vascular monitoring device (intervention group, n=25) against those with standard care clinical observation (control group, n=25). Descriptive statistics will be used to summarise the results that will assess the vascular monitoring capability of implantable Doppler probe in the early postoperative period of kidney transplant patients. The results will provide estimates for surgical outcomes essential to inform the sample size calculation for the definitive study. Information related to the fluency of research methods, availability of research resources, management support, potential challenges faced during the fRCT will be compiled to generate realistic estimates of important parameters for the definitive study. The results will be following the CONSORT updated guidelines for reporting feasibility studies.

Qualitative semi-structured interviews of stakeholders (n=12) recruited by purposive sampling will be conducted to explore their experiences of participating in the study, acquire suggestions regarding application of implantable Doppler probe monitoring, and the post implantation patient care. All interviews will be audio-recorded with verbatim transcription. Data will be analysed following the six-phase guide to doing thematic analysis in the NVivo software. The results will be reported in accordance with the consolidated criteria for reporting qualitative research (COREQ) checklist.

IMPACT It is anticipated that this study will also elaborate on a possible role of implantable Doppler probe monitoring to improve kidney transplant patient safety, graft survival, service quality improvement, and financial savings in the NHS.

DETAILED DESCRIPTION:
AIM:

To evaluate the usefulness of an implantable continuous vascular monitoring device in kidney transplant surgery and to inform the protocol development of a definitive planned RCT.

OBJECTIVES

Feasibility RCT OBJECTIVE 1 To assess the capability of the implantable vascular monitoring device in the early postoperative period of kidney transplant patients.

OBJECTIVE 2 To assess the research methods used to compare vascular monitoring device with the standard care and to estimate surgical outcome measures essential to inform the sample size calculation for the definitive planned RCT.

OBJECTIVE 3 To assess the availability of research resources, management support, potential barriers and challenges for the definitive planned RCT.

EMBEDDED QUALITATIVE STUDY OBJECTIVE 4 To assess the acceptability of vascular monitoring device in clinical practice and get suggestions on the protocol development of the definitive planned RCT TRIAL DESIGN Mixed methodology two-arm feasibility randomised controlled trial with an embedded qualitative study.

RECRUITMENT The participants will be recruited from the patients undergoing kidney transplant surgery at Southwest transplant centre, UHPNT. The chief investigator will recruit the eligible participants and obtain their consent for the study. The normal care pathway followed at our transplant unit is designed in line with the unpredictable nature of the speciality. The investigators are offered organs by NHS Blood and Transplant (NHSBT) from deceased donors with a notice period of 12-14 hours. The kidney transplant recipient is admitted to the hospital about 8-10 hours before the surgery. The patient is prepared and consented to surgery during this interval. The patient is then moved to the operation theatre for transplantation. After surgery, the patient is transferred to the renal ward for postoperative care. All patients receive standard care clinical observation to monitor their graft function. In addition to the standard care clinical observation, the clinician looking after the patients may request additional departmental ultrasound scans in the first 72 hours depending on the graft function and the condition of the kidney transplant recipient.

There will be no difference in the recruitment process, consent, and the postoperative care of kidney transplant patients with the monitoring device or with the standard care clinical observation.

TRIAL PARTICIPANTS The participants of the study will consist of the patients who will have kidney transplant surgery with or without the implantable vascular monitoring device during the study duration at the Southwest transplant centre UHPNT.

TRIAL SETTINGS Southwest transplant centre, University Hospitals of Plymouth NHS trust. DURATION OF THE STUDY 24 months SAMPLE SIZE The sample size is chosen based on the practicalities of conducting a feasibility study. The sample size is a realistic recruitment figure for 24 months based on a recent retrospective study conducted at the Southwest transplant centre leading to this research project. The data suggested that about 65-70 kidney transplants were performed annually in our unit. The randomised controlled feasibility trial aims to recruit 50 kidney transplant patients within a 24-month period; 25 in intervention group and 25 in control group. In this study, the investigators propose to attach an implantable continuous vascular monitoring device to half (i.e. 25) of the kidney transplant patients (intervention Group) during their surgery. Postoperatively, these patients will receive graft surveillance by the monitoring device in addition to the standard care clinical observation. The other half (i.e. 25) of the kidney transplant patients (control Group) will receive the standard care clinical observation.

CONSENT The chief investigator (CI) will inform the patients about the study and invite them to participate. Consent to enter the study will be sought from each participant only after a full explanation of the study. An information leaflet will also be offered. A duly signed informed consent form will be obtained from patients that agree to participate in the study.

RANDOMISATION The patients who consent to participate in the study will be randomised into two groups (i.e. intervention and control) by a secure online computer sequence generator system (https://www.randomizer.org/#randomize). Randomisation will be completed in a 1:1 ratio using random permuted blocks.

The patients allotted to the Intervention group will have kidney transplants with the implantable continuous vascular monitoring device while those allotted to the Control group will have kidney transplants with standard care clinical observation (i.e. without implantable continuous vascular monitoring device).

TRIAL ARMS INTERVENTION GROUP (KIDNEY TRANSPLANT PATIENTS WITH THE IMPLANTABLE CONTINUOUS VASCULAR MONITORING DEVICE) The intervention that is intended to be investigated is the implantable continuous vascular monitoring device manufactured by COOK Medical Company. Its principle intended use is continuous monitoring of the graft perfusion (i.e. transplanted kidney) for the first 72 hours postoperatively. The kidney transplant patients in the intervention group will receive implantable continuous vascular monitoring device surveillance for the first 72 hours in addition to the standard care clinical observation as part of their postoperative care. The device will be removed after 72 hours.

CONTROL GROUP (KIDNEY TRANSPLANT PATIENTS WITH STANDARD CARE CLINICAL OBSERVATION):

The kidney transplant patients in this group will receive the standard care clinical observation as part of their postoperative care. Their graft will be monitored postoperatively by the standard care clinical observation as per the NHS protocol.

BLINDING Blinding of the participants (kidney transplant patients) to the outcome of the randomisation will not be possible due to the nature of the intervention. Similarly, the healthcare professionals (clinicians and nurses) taking care of the patients and collecting the data postoperatively cannot be blinded.

DATA COLLECTION Data collection will take place in the immediate period after the kidney transplant in recovery, at 24, 48, and 72 hours postoperatively in the ward and at the three-monthly postoperative clinic visit.

The data will be collected prospectively and independently for both groups over a two year period. Data collection may culminate earlier if the required sample size is achieved. It will include participant's demographic characteristics and the outcomes that will be measured to achieve the respective objectives of the study.

INTENTION TO TREAT ANALYSIS The data of the participants who will be randomised into the two groups (i.e. Intervention Group and Control Group) will be summarised separately in their respective groups.

DATA ANALYSIS It is inappropriate to use inferential statistics in feasibility study data to formally test the effectiveness of an intervention. Data analyses using descriptive statistics will be performed in IBM SPSS version 25.0. The means and standard deviations will be considered as the representative value of the continuous variables (i.e. participant's demographic characteristics). The categorical variables (i.e. surgical outcomes) will be expressed by frequency distributions (percentages) and elaborated using tables and graphs.

The participant's demographic or baseline characteristics in both groups will be summarised separately using descriptive statistics. The numerical data for both groups will be compared in the tabular form to demonstrate whether or whether not the participant's baseline characteristics in the Intervention and Control groups are identical.

The outcomes for each objective in both groups (i.e. intervention and control) will be summarised using descriptive statistics. The numerical data from both groups will be compared to describe the feasibility of the intervention and generate realistic estimates of important parameters for the definitive multi-centre RCT.

EMBEDDED QUALITATIVE STUDY AIM This component of the trial is aimed at exploring the experiences (receiving/delivering the intervention) and suggestions of the stakeholders on participating in the study.

OBJECTIVE To assess the acceptability of vascular monitoring device in clinical practice and to acquire suggestions and innovative ideas of the stakeholders on refining the design of definitive RCT, functioning of the implantable vascular monitoring device, and improving postoperative patient care.

STUDY DESIGN An exploratory inductive approach will be used with the qualitative study design of phenomenology. Semi-structured interviews with open-ended questions will be used.

PARTICIPANTS To ensure the selection of information-rich cases and to attain an all-around perspective consistent with the aim of this study, a purposeful sampling consisting of participants from all groups involved with the device will be done. The participants of the study must have experience with the vascular monitoring device and will be selected according to whoever is on-call on the day of kidney transplant according to the clinicians and nurse's duty rotation plan. They will comprise four clinicians, four nurses, and four kidney transplant patients. Maximum sample number (12) is described however; recruitment will be discontinued early if theoretical saturation is attained.

Consent for the interview and further correspondence for member-checking will be obtained at the time.

DATA COLLECTION The qualitative study will consist of semi-structured interviews with open-ended questions and conducted in line with the NIHR's instructions laid out in the health and social care research handbook for researchers. The interview guide used will compromise key steps like introduction, a brief description of the proposed study, explanation of the purpose of the study, consent, and interview questions which will be aided by probing questions if further elaboration is required.

The duration of the interviews will last 40-45 minutes. The interview proceedings will be audio recorded with the participant's consent and will be deleted following transcription. The participants will be informed that any quotes used in the report would be pseudonymised and kept strictly confidential. Field notes will be taken during all interview sessions to ensure the richness of data.

Interviews will be conducted in the kidney ward, which is selected to enable participants to relax and open up in their routine setup. The privacy of the interviews will be maintained to allow participant anonymity and will take place during the lunch break to avoid distractions from the clinical commitments.

DATA ANALYSIS Thematic analysis will be performed in NVivo 12 qualitative analysis program. The chief investigator has a theoretical interest in the device. To reduce the potential for interviewer bias, the thematic analysis will be conducted by the inductive approach of data-driven identification of themes. Since all participants will have experience with the device, the thematic analysis will be done at the latent level to identify the underlying ideas and assumptions. Data extracts will be coded and categorised into themes, following the six-phase guide to doing thematic analysis.

The result of this study will be reported in accordance with the Consolidated criteria for reporting qualitative research (COREQ) checklist.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will have deceased or living kidney donor transplants
2. Patients aged 18 years or above.
3. Patients able and willing to comply with the trial requirements

Exclusion Criteria:

1. Patients who will have a kidney transplant with more than two arteries (evident at the time of surgery).
2. Patients below 18 years of age.
3. Patients lacking capacity or unwilling to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
OBJECTIVE 1: To assess the capability of vascular monitoring device in the early postoperative care of kidney transplant patients This objective will be achieved in the feasibility randomised controlled trial. | 12 weeks
  OUTCOME MEASURES FOR OBJECTIVE 1:
  The following outcomes in both the intervention and control groups will be recorded and compared to measure the objective 1.
  1. The number of early vascular complications identified in each group (measured as numerical number i.e.,1,2,3 etc).
  2. The number of departmental ultrasound scans requested in the first 24, 48, and 72 hours postoperatively in each participant (measured as numerical number i.e.,1,2,3 etc).
  3. The number of grafts lost due to vascular complications in each group (measured as numerical number i.e.,1,2,3 etc).
OBJECTIVE 2: To assess the research methods used in this feasibility randomised for the definitive planned randomised controlled study This objective will be achieved in the feasibility randomised controlled trial. | 12 weeks
  OUTCOME MEASURES FOR OBJECTIVE 2:
  The suitability of the following research processes used in the study will be estimated. Any difficulties or shortcomings encountered will be highlighted.
  1. Difficulties encountered with eligibility criteria and recruitment process (measured as a binary variable i.e., Yes or No).
  2. Difficulties encountered with randomisation or allocation concealment (measured as a binary variable i.e., Yes or No).
  3. Difficulties encountered with retention/follow-up/compliance of participants (measured as a binary variable i.e., Yes or No).
  4. Variation or fidelity encountered in the delivery of the intervention marked against a fidelity checklist (measured as a binary variable
  i.e., Yes or No)
OBJECTIVE 3: To assess the availability of research resources, management support, potential barriers and challenges for the definitive planned future RCT. This objective will be achieved in the feasibility randomised controlled trial. | 12 weeks
  OUTCOME MEASURES FOR OBJECTIVE 3:
  The availability of the following research resources in this study will be recorded. Any shortcomings or non-availability of resources encountered will be highlighted.
  1. Availability of participant documentation (i.e., participant information sheet, consent form, data collection sheet) (measured as a binary variable i.e., Yes or No).
  2. Availability of medical equipment and healthcare staff in the host centre required to handle the number of participants and the research procedures (measured as a binary variable i.e., Yes or No).
  3. Availability of technological capacity for communication and adequate software to randomise, record, process, and store research data (measured as a binary variable i.e., Yes or No).
  4. Availability of management support for the research project and back up plans for any extenuating circumstances (measured as a binary variable i.e., Yes or No).
Objective 4: To assess the acceptability of the ID probe blood flow monitoring device in clinical practice and get suggestions for the definitive planned future RCT. This objective will be achieved by the embedded qualitative study | 12 weeks
  OUTCOME MEASURES FOR OBJECTIVE 4:
  The acceptability of the intervention in clinical practice will be assessed by conducting the thematic analysis of the views and experiences of stake holders (clinicians, transplant surgeons, nurses, and kidney transplant patients with the experience of receiving/delivering the intervention and participating in the study) obtained by qualitative interviews with open ended questions. Furthermore, suggestions to improve the design of the definitive planned future RCT, functioning of the ID probe blood flow monitoring device, or any aspect of postoperative patient care will also be acquired.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fern, PhD, Study Director — Peninsula Medical School (Faculty of Health), University of Plymouth; M Shahzar Malik, MClinRes, Principal Investigator — University Hospitals Plymouth NHS Trust; Kris Houlberg, PhD, Study Chair — University Hospitals Plymouth NHS Trust; Aled Jones, PhD, Study Director — Head of School of Nursing and Midwifery, University of Plymouth
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
DATA MANAGEMENT PLAN A data management plan for this study was prepared under the University of Plymouth's information governance Policy, the UK General Data Protection Regulation (GDPR-2018), and Good Clinical Practice (GCP). It consists of a complete plan for data protection, retention, and erasure after 10 years.
  During the data collection, patient information in fRCT and embedded qualitative study will be pseudonymised and kept strictly confidential by the CI using a unique anonymised code, ensuring it does not contain any patient identifiers. The renal database (Vital Data) will be used for the information extraction and is password protected present only on the Trust intranet.
  All data protection measures will be undertaken to maintain the confidentiality of the participants. The official NHS email address will be used for the transfer of any pseudonymised information if required.

REFERENCES:
- [Result] Schmulder A, Gur E, Zaretski A. Eight-year experience of the Cook-Swartz Doppler in free-flap operations: microsurgical and reexploration results with regard to a wide spectrum of surgeries. Microsurgery. 2011 Jan;31(1):1-6. doi: 10.1002/micr.20816. PMID 20683856
- [Result] Hakim DN, Nader MA, Sood A, Kandilis A, Hakim NS. Rescue of Transplanted Kidney Thanks to an Implantable Doppler Probe: Is This the Future? Exp Clin Transplant. 2016 Aug;14(4):454-5. doi: 10.6002/ect.2014.0135. Epub 2014 Oct 21. PMID 25343411
- [Result] Lenz Y, Gross R, Penna V, Bannasch H, Stark GB, Eisenhardt SU. Evaluation of the Implantable Doppler Probe for Free Flap Monitoring in Lower Limb Reconstruction. J Reconstr Microsurg. 2018 Mar;34(3):218-226. doi: 10.1055/s-0037-1608628. Epub 2017 Nov 27. PMID 29179224
- [Result] Chang TY, Lee YC, Lin YC, Wong ST, Hsueh YY, Kuo YL, Shieh SJ, Lee JW. Implantable Doppler Probes for Postoperatively Monitoring Free Flaps: Efficacy. A Systematic Review and Meta-analysis. Plast Reconstr Surg Glob Open. 2016 Nov 28;4(11):e1099. doi: 10.1097/GOX.0000000000001099. eCollection 2016 Nov. PMID 27975015
- [Result] Vasant Kulkarni S, Rao PP, Naidu CS, Pathak N, Singh AK. Evaluation of implantable Doppler probe continuous monitoring of hepatic artery anastomosis after liver transplantation. Med J Armed Forces India. 2021 Jul;77(3):349-354. doi: 10.1016/j.mjafi.2020.03.012. Epub 2020 Jun 3. PMID 34305290
- [Result] Poder TG, Fortier PH. Implantable Doppler in monitoring free flaps: a cost-effectiveness analysis based on a systematic review of the literature. Eur Ann Otorhinolaryngol Head Neck Dis. 2013 Apr;130(2):79-85. doi: 10.1016/j.anorl.2012.07.003. Epub 2012 Nov 23. PMID 23182889
- [Result] Crane J, Hakim N. The use of an implantable Doppler flow probe in kidney transplantation: first report in the literature. Exp Clin Transplant. 2011 Apr;9(2):118-20. PMID 21453229
- [Result] de Jong KP, Bekker J, van Laarhoven S, Ploem S, van Rheenen PF, Albers MJ, van der Hilst CS, Groen H. Implantable continuous Doppler monitoring device for detection of hepatic artery thrombosis after liver transplantation. Transplantation. 2012 Nov 15;94(9):958-64. doi: 10.1097/TP.0b013e318269e6ad. PMID 23037006

DOCUMENTS (3):
  • Study Protocol (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT05634863/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT05634863/SAP_001.pdf
  • Informed Consent Form (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT05634863/ICF_002.pdf